CLINICAL TRIAL: NCT04065035
Title: A Double-Blind Split-Body Placebo-Controlled Clinical Study to Evaluate the Efficacy of a Cosmetic Product for Arm Firming
Brief Title: A Clinical Study to Evaluate Efficacy and Tolerability of a Cosmetic Product for Arm Firming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: Stephens & Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C18-D134
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Photodamaged Skin; Skin Care
Keywords: Body; moisturizer; Firming
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Split Body, randomized, and placebo controlled
Who Masked: Participant, Investigator
Masking Description: Prior to the start of the study, Stephens will generate 2 randomization lists (1 for biopsy subjects and 1 for non-biopsy subjects) to establish treatment assignment to 1 arm (left or right) with the other arm untreated (receiving a placebo). Each list will first be created by concatenating blocks of size of 4 subjects, 2 with left arm treated/right arm untreated and 2 with right arm treated/left arm untreated. The lists will then be randomized by variables from 2 independent uniform distributions: 1 to randomize subjects within block and 1 to randomize blocks. After the randomization lists are created, treatment arm will be assigned to each subject number accordingly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Firming Body Moisturizer (Active Comparator): Oil-in-water emulsion base containing emollients, botanical extracts, peptides, antioxidants, prebiotics, and modified theophylline ingredients.
  Interventions: Other: Topical Body Firming Moisturizer; Other: Body Cleanser; Other: Sunscreen
- Placebo Moisturizer (Placebo Comparator): Oil-in-water emulsion base containing emollients.
  Interventions: Other: Body Cleanser; Other: Sunscreen; Other: Placebo Moisturizer

INTERVENTIONS:
Other: Topical Body Firming Moisturizer — Moisturizer composed of a patent-pending blend of botanical extracts, bioavailable peptides, antioxidants, and a prebiotic innovation
  Arms: Topical Firming Body Moisturizer
Other: Body Cleanser — Body cleanser to be used by study participants
  Other Names: Dove Sensitive Skin Nourishing Body Wash
Other: Sunscreen — Sunscreen to be applied after application of moisturizer
  Other Names: Neutrogena® Ultra Sheer® Dry-Touch Sunscreen Broad Spectrum Sunscreen Protection Factor 55
Other: Placebo Moisturizer — Placebo moisturizer is the vehicle control of the topical body firming moisturizer
  Arms: Placebo Moisturizer

SUMMARY:
This single-center, split-body, double-blind, randomized, controlled clinical trial was conducted to assess the efficacy and tolerance of a topical firming body moisturizer when used over the course of 12 weeks by women with mild to moderate sagging, crepey skin, and overall photodamage on the upper arms. A total of 40 subjects completed study participation which included 10 subjects in the biopsy subgroup.

DETAILED DESCRIPTION:
This single-center, split-body, double-blind, randomized, controlled clinical trial is being conducted to assess the efficacy and tolerance of the topical firming body moisturizer when used over the course of 12 weeks by women with mild to moderate sagging, crepey skin, and overall photodamage on the upper arms.

Efficacy and tolerance will be assessed through clinical grading at baseline and weeks 4, 8, and 12. Efficacy will also be assessed through Corneometer and upper arm circumference measurements at baseline and weeks 4, 8, and 12, and Cutometer and Ultrasound measurements at baseline and weeks 8 and 12. Self-assessment questionnaires will be completed at baseline and week 12. Digital images will be taken at baseline and weeks 4, 8, and 12. Vectra H2 3D images will be taken at baseline and weeks 8 and 12. BMI will be measured at baseline and weeks 8 and 12. Biopsies will be collected from a subgroup of at least 10 subjects at baseline and week 12 (two biopsies on each arm at each time point; total of 8 per biopsy subject).

A total of 40 subjects completed study participation which included 10 subjects in the biopsy subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 40 and 60 years
* Mild to moderate skin crepiness upper arm region
* Mild to moderate sagging skin upper arm region
* Mild to moderate overall photodamage upper arm region
* Willing to maintain their body weight within +/- 6.5 pounds

Exclusion Criteria:

* Diagnosed with known allergies to skin care products
* Who have had massive weight loss
* Who have undergone liposuction and/or weight loss surgery in the last 5 years.
* Who are nursing
* Who are pregnant
* History of skin cancer within the past 5 years.
* Having a health condition
* Having a history of immunosuppression/immune deficiency disorders
* Currently using oral or systemic immunosuppressive medications and biologics
* Currently using or having regularly used corticosteroids
* Having a disease such as asthma
* Having started a long-term medication within the last 2 months.
* Who started hormone replacement therapies (HRT)
* Having had brachioplasty (upper arm lift);
* Having liposuction
* Having cryolipolysis
* Having undergone a weight-loss diet or exercise habit change in the last 3 months or planning to start either during the study.
* Having used any of the indicated products or had any of the listed procedures on the upper arms within the indicated time frame prior to the study start date.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Skin Crepiness Score | 12 weeks
  Investigator assessed the participants' skin crepiness using a 10-point scale where none 0 = skin appears smooth with no crinkling to severe 9 = prominent, extensive crinkly texture at baseline, week 4, 8, and 12. A decrease in score indicates improvement.
Change from Baseline in Skin Elasticity Score | 12 weeks
  Investigator assessed the participants' skin elasticity using a 10-point scale where none 0 = skin feels toned, dense and resilient to severe 9 = skin feels pliable, thin and nonresilient at baseline, week 8 and 12. A decrease in score indicates improvement.
Change from Baseline in Skin Firmness Score | 12 weeks
  Investigator assessed the participants' skin firmness using a 10-point scale where none 0 = skin appears very firm and feels thick to severe 9 = loose-appearing skin with poor stretch properties at baseline, week 8 and 12. A decrease in score indicates improvement.
Change from Baseline in Skin Sagging Score | 12 weeks
  Investigator assessed the participants' skin sagging using a 10-point scale where none 0 = no sagging, upper arm shows tight, lifted appearance to severe 9 = upper arm shows extreme sagging appearance at baseline, week 8 and 12. A decrease in score indicates improvement.
Change from Baseline in Skin Roughness (Visual) Score | 12 weeks
  Investigator assessed the participants' skin roughness (visual) using a 10-point scale where none 0 = smooth skin appearance, no roughness to severe 9 = pronounced reduction in skin smoothness appearance at baseline, week 4. 8, and 12. A decrease in score indicates improvement.
Change from Baseline in Skin Roughness (Tactile) Score | 12 weeks
  Investigator assessed the participants' skin roughness (tactile) using a 10-point scale where none 0 = no palpable skin roughness, drag or surface bumps to severe 9 = significantly palpable skin roughness, drag, and surface bumps at baseline, week 4, 8 and 12. A decrease in score indicates improvement.
Change from Baseline in Overall Photodamage Score | 12 weeks
  Investigator assessed the participants' overall photodamage using a 10-point scale where none 0 = none or minimal visual evidence of photodamaged skin to severe 9 = severe photodamaged skin at baseline, week 8 and 12. A decrease in score indicates improvement.
Change from Baseline in Evenness of Skin Tone Score | 12 weeks
  Investigator assessed the participants' evenness of skin tone using a 10-point scale where none 0 = even skin color, no observable hyperpigmentation to severe 9 = significant detectable hyperpigmentation appearance at baseline, week 8 and 12. A decrease in score indicates improvement.
Change from Baseline in Evenness of Skin Redness Score | 12 weeks
  Investigator assessed the participants' evenness of skin redness using a 10-point scale where none 0 = even skin tone to severe 9 = pronounced areas of redness at baseline, week 4, 8, and 12. A decrease in score indicates improvement.
Change from Baseline in Objective Erythema Parameters | 12 weeks
  Investigator assessed the participants' signs of erythema using a 4-point scale where none 0 = no erythema to severe 4 = marked redness at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Objective Edema Parameters | 12 weeks
  Investigator assessed the participants' signs of edema using a 4-point scale where none 0 = no edema or swelling to severe 4 = marked edema at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Objective Dryness Parameters | 12 weeks
  Investigator assessed the participants' signs of dryness using a 4-point scale where none 0 = no dryness to severe 4 = marked dryness at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Objective Peeling Parameters | 12 weeks
  Investigator assessed the participants' signs of peeling using a 4-point scale where none 0 = no peeling to severe 4 = marked peeling at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Subjective Burning Parameters | 12 weeks
  Participants assessed signs of burning using a 4-point scale where none 0 = no burning to severe 4 = hot burning sensation at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Subjective Stinging Parameters | 12 weeks
  Participants assessed signs of stinging using a 4-point scale where none 0 = no stinging to severe 4 = marked stinging sensation at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Subjective Itching Parameters | 12 weeks
  Participants assessed signs of itching using a 4-point scale where none 0 = no itching to severe 4 = marked itching sensation at baseline and week 12. A decrease in score indicates improvement.
Change from Baseline in Subjective Tingling Parameters | 12 weeks
  Participants assessed signs of tingling using a 4-point scale where none 0 = no tingling to severe 4 = marked tingling sensation at baseline and week 12. A decrease in score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Jiang, PhD, Principal Investigator — Thomas J. Stephens & Associates, Inc
Locations (1):
- Stephens and Associates, Richardson, Texas, United States